CLINICAL TRIAL: NCT02974270
Title: Analysis of Body Mass Index in Central Precocious Puberty(CPP) Patients Treated With Leuprolide Acetate
Brief Title: Analysis of Body Mass Index in Central Precocious Puberty Patients Treated With Leuprolide Acetate
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Woo Ko, MD, PhD, Kyungpook National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IISR-2014-100760
Record Dates: First submitted 2016-05-19; First posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Precocious Puberty, Central
MeSH Terms: conditions — Puberty, Precocious | interventions — Leuprolide

ARMS (1):
- Leuprolide acetate (Experimental)
  Interventions: Drug: Leuprolide

INTERVENTIONS:
Drug: Leuprolide

SUMMARY:
Analysis of body mass index in Central Precocious Puberty patients treated with leuprolide acetate

ELIGIBILITY:
Inclusion Criteria:

1. Child diagnosed with CPP who has a peak-stimulated Lutenizing Hormone(LH) concentration over 5 IU/liter before initiation of therapy
2. Chronological age(CA) at the appearance of pubertal changes less than 8 years in girls and less than 9 years in boys.
3. Tanner stage ≥2
4. Advanced bone age (Bone Age/Chronological Age >1.1)
5. Able to have the signed written informed consent provided by the patients' parents or legal guardians prior to any study-related procedures

Exclusion Criteria:

1. Patient with a peripheral precocious puberty: extrapituitary secretion of gonadotropins or gonadotropin-independent gonadal or adrenal sex steroids secretion
2. Patient with a cerebral tumor requiring a neurosurgery or cerebral irradiation known chronic disease of underlying medical condition
3. Currently on or planning growth hormone treatment
4. Previous Gonadotropin-Releasing Hormone agonist treatment
5. Any patient who in opinion of the investigator should not participate in the study

Max Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Body Mass Index Standard Deviation Score for Chronological Age at 6 months | 6 months

SECONDARY OUTCOMES:
Change from baseline Body Mass Index Standard Deviation Score for Chronological Age at 3 months | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cheol Woo Ko, Daegu, South Korea